CLINICAL TRIAL: NCT01525108
Title: A Home-based Blood Pressure Measurement Program in Hypertensive Patients to Promote Medications Adherence and Blood Pressure Status.
Brief Title: A Home-based Blood Pressure Monitoring Program to Promote Better Management of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Research Center for Rational Use of Drugs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90-04-156-15281
Record Dates: First submitted 2012-01-30; First posted 2012-02-02 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Hypertension
Keywords: Medication adherence; Blood pressure; Home-based blood pressure measurement; Blood Pressure Determination; Blood Pressure Monitors; Blood Pressure Monitoring, Ambulatory
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-based blood pressure monitoring (Experimental)
  Interventions: Behavioral: Self monitoring of blood pressure
- Usual care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Self monitoring of blood pressure — Electronic blood pressure device is provided for patients and he/she will be trained to measure blood pressure at home once daily(same time each day). A logbook is also provided to document the daily blood pressure level.
  Arms: Home-based blood pressure monitoring
Other: Usual Care — Four visits to the physician's office at 4th, 12th, 24th week in the study period with usual advice giving practice of the staff. At the end of the trial period, an electronic blood pressure device will be given to each patient in this arm.
  Arms: Usual care

SUMMARY:
In this study the investigators aim to evaluate the effect of home-based blood pressure measurement with an electronic device on medication adherence and blood pressure control.

DETAILED DESCRIPTION:
Adherence to treatment is disappointingly low among patients with chronic health disorders especially after 6 month of initiating drug therapy. In hypertensive patients , as reported by WHO, 50% of non-adherence could be expected. Poor adherence to anti hypertensive medications results in increased morbidity, mortality and costs. One of the reasons that could implicate medications adherence can be attributed to seeing no physical sign of better controlling blood pressure. Self monitoring of blood pressure at home has been reported to improve patients adherence to their medications.

This study is a 2-arm randomized controlled trial. The investigators aim to evaluate the effect of home-based blood pressure measurement with an electronic device on medication adherence and blood pressure status.

One hundred ninety six hypertensive patients aged at least 18 years old are recruited in an ambulatory care setting and are evenly allocated to the study arms with balanced-block telephone randomization.

Appropriate medication is prescribed as preferred by the cardiologist (single daily dose medicines are recommended). Patients in both arms are followed for 24 weeks, each will be visited by the cardiologist four times during the study period. In each visit, patients' blood pressure will be measured twice by a nurse in the office.

In the intervention arm, electronic blood pressure device is provided for each patient and he/she will be trained to measure blood pressure at home once daily (same time each day). A logbook is also provided to document the daily blood pressure level.

Primary outcome of the study is the blood pressure measured at each office visit overtime. Medication adherence is measured by pill count method as the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients older than 18
* Patients newly diagnosed as hypertension stage 1
* Patients previously on antihypertensive treatment but uncontrolled hypertension
* Patients not possessing electronic self blood pressure measurement device
* Patients with functional ability to use the device

Exclusion Criteria:

* Patients requiring two or more antihypertensive drugs at the start of the study
* Patients with secondary hypertension
* Patients cardiovascular comorbidities and other interfering medical conditions
* Patients with drug contraindication or documented drug allergy
* Patients with serum creatinine > 150 microliters

Withdrawal criteria:

* Inadequate therapeutic effect requiring an increase of more than 20% in pre-established number of visits
* Emergence of adverse drug reactions requiring cessation of medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure-24 weeks | Change from baseline(at the point of recruiting) blood pressure at 24 weeks.
  Blood pressure is measured twice by trained nurses using hand-cuff device at the physician office. (in Hg millimeter)

SECONDARY OUTCOMES:
Medication adherence-4 weeks | Change from baseline(at the point of recruiting) medication adherence at 4 weeks
Blood pressure- 4 weeks | Change from baseline(at the point of recruiting) blood pressure at 4 weeks.
Blood pressure- 12 weeks | Change from baseline(at the point of recruiting) blood pressure at 12 weeks.
Medication adherence- 12 weeks | Change from baseline(at the point of recruiting) medication adherence at 12 weeks
Medication adherence-24 weeks | Change from baseline(at the point of recruiting) medication adherence at 24 weeks
  Pill count method is employed. At the time of each office visit, patients bring their medications with themselves and the researcher counts the unused pills. Adherence is calculated as percentage of the pills used during previous weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kheirollah Gholami, M.Sc,PharmD, Study Chair — Tehran University of Medical Sciences; Zahra Jahangard-Rafsanjani, PharmD, Study Director — Tehran University of Medical Sciences; Arash Rashidian, M.D, Ph.D, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Dr Mohagheghi's Office, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Hosseininasab M, Jahangard-Rafsanjani Z, Mohagheghi A, Sarayani A, Rashidian A, Javadi M, Ahmadvand A, Hadjibabaie M, Gholami K. Self-monitoring of blood pressure for improving adherence to antihypertensive medicines and blood pressure control: a randomized controlled trial. Am J Hypertens. 2014 Nov;27(11):1339-45. doi: 10.1093/ajh/hpu062. Epub 2014 Apr 26. PMID 24771706